CLINICAL TRIAL: NCT01578668
Title: Phase 2 Study of Erlotinib Plus Pemetrexed/Cisplatin Treating Lung Adenocarcinoma With Brain Metastases
Brief Title: Erlotinib Plus Pemetrexed to Treat Lung Adenocarcinoma With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Haihong Yang, MD, Pricipal investigator, The first affiliated hospital of Guangzhou MC, Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZTO1201
Record Dates: First submitted 2012-04-11; First posted 2012-04-17 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Lung Adenocarcinoma; Brain Metastases
Keywords: lung adenocarcinoma; brain metastases; erlotinib; pemetrexed
MeSH Terms: conditions — Adenocarcinoma of Lung; Brain Neoplasms | interventions — Erlotinib Hydrochloride; Pemetrexed; Cisplatin; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib, pemetrexed, cisplatin (Experimental)
  Interventions: Drug: erlotinib; Drug: pemetrexed; Drug: cisplatin
- erlotinib (Experimental)
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — 150 mg given orally (po), daily (QD), starting on the 4th day of each cycle, ending on the 21th day before the next cycle, and until disease PD
  Other Names: Tarceva
  Arms: Erlotinib, pemetrexed, cisplatin
Drug: pemetrexed — 500 mg/m² intravenous (iv) over 15 minutes on the first day of each 21-day cycle until disease progression (PD) or unacceptable toxicity or no more than 6 cycles
  Other Names: ALIMTA
  Arms: Erlotinib, pemetrexed, cisplatin
Drug: cisplatin — cisplatin 20mg/m² iv on the 1st-3rd day (if PS<2) or 30 mg iv on the 1st-2nd day (if PS=2 or 3)of each cycle until PD or unacceptable toxicity or no more than 6 cycles
  Other Names: platinum
  Arms: Erlotinib, pemetrexed, cisplatin
Drug: erlotinib — 150 mg given orally (po), daily (QD), starting on the first day of the first cycle
  Other Names: Tarceva
  Arms: erlotinib

SUMMARY:
The purpose of this study is to determine whether erlotinib plus pemetrexed, cisplatin are effective and safe in treating lung adenocarcinoma with brain metastases.

DETAILED DESCRIPTION:
Non-small lung cancer (NSCLC) is the leading cause of death in the world. Brain metastases are a frequent complication of NSCLC, especially in lung adenocarcinoma. 30-50% or more these patients will develop brain metastases at first time or during the treatment. Limited treatment options, whole brain radiotherapy (WBRT) combined with or without stereotactic radiosurgery (SRS) as the primary treatment approach, are available for brain metastases patients with poor survival. So the availability of effective therapies are therefore of great importance. Currently, two agents (erlotinib and pemetrexed) are reported more effective in lung adenocarcinoma patients with brain metastases. The heterogeneity of NSCLC tumors provides a strong rationale for using combination therapy with targeted agents that have different mechanisms of action, moreover different combination offering synergistic effects. So we investigate if erlotinib plus pemetrexed, cisplatin are effective and safe in treating lung adenocarcinoma with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of lung adenocarcinoma histology with brain metastases
2. 18 years or older
3. Eastern Cooperative Oncology Group (ECOG) Performance Status no more than 3 (poor PS caused by neurological symptom)
4. Appraisable intracranial disease, the presence of at least one lesion, and the longest diameter > 5 mm by brain MRI
5. Haemoglobin 10.0 g/dl, Absolute neutrophil count (ANC) 1.5^9/L, platelets 100 x 10^9/L
6. Total bilirubin 1.5 x upper limit of normal (ULN)
7. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases
8. Creatinine clearance 60ml/min (calculated according to Cockcroft-gault formula)
9. If received brain radiotherapy, patients included at least 8 weeks after the end of radiotherapy.

Exclusion Criteria:

1. Mixed non-adenocarcinoma cell lung cancer histology
2. Previous treatment with pemetrexed or tarceva
3. Be allergic to pemetrexed or tarceva

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The objective response rate of brain metastases | Patients will be followed for an expected average of 6 weeks

SECONDARY OUTCOMES:
The disease control response rate of disease | Patients will be followed for an expected average of 6 weeks
Progression-free survival of patients | 2 years after first treatment
Number of participants with adverse events as a measure of safety | 2 years after first treatment
Overall survival of patients | 3 years after the first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Haihong Yang, Dr., Principal Investigator — The first affiliated hospital of Guangzhou MC
Locations (1):
- The first affiliated hospital of Guangzhou MC, Guangzhou, Guangdong, China